CLINICAL TRIAL: NCT07038538
Title: Evidence-based Practice in the Management of Gastric Tube Placement in Children: A Multicenter Quality Improvement Project
Brief Title: Evidence-based Practice in the Management of Gastric Tube Placement in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Guangzhou Women and Children's Medical Center (Other); Children's Hospital of Chongqing Medical University (Other); Gansu Provincial Maternity and Child-care Hospital/Gansu Provincial Central Hospital (Unknown); Hunan Children's Hospital (Other Government); Children's Hospital, Zhejiang University School of Medicine (Unknown); The First Hospital of Jilin University (Other); Jinan Maternity and Child Health Care Hospital (Unknown); Henan Provincial People's Hospital (Other); Shengjing Hospital (Other); Shenzhen Children's Hospital (Other Government); Kunming Children's Hospital (Other); Tongji Hospital (Other); Anhui Provincial Children's Hospital (Other); Children's Hospital of Nanjing Medical University (Other); Children's Hospital of Soochow University (Other); The First People's Hospital of Urumqi （Urumqi Children's Hospital) (Unknown); Peking University First Hospital (Other); Qingdao Women and Children's Hospital (Unknown); Capital Center for Children's Health,Capital Medical University (Unknown); Beijing Children's Hospital (Other); West China Second University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHFudanU1110
Record Dates: First submitted 2024-11-11; First posted 2025-06-26 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hospitalized Children; Nursing; Enteral Nutrition Therapy
Keywords: Quality Improvement; Before-and-After Comparison; Cognitive and behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evidence-based gastric tube placement (Experimental): To implement gastric tube placement management scheme, then observe the continuous changes.
  Interventions: Behavioral: Evidence-based gastric placement

INTERVENTIONS:
Behavioral: Evidence-based gastric placement — Establish an enteral nutrition management team and develop standardized procedures through a quality improvement project. Conduct a 3-month quality improvement initiative, during which regular training sessions will be provided to nurses on gastrointestinal tube placement and maintenance. These training sessions will include various formats such as lectures, group discussions, operational demonstrations, and scenario simulations, along with regular reviews of practical issues.

SUMMARY:
This multi-center quality improvement project aims to enhance gastric tube placement practices for children by systematically reviewing the latest evidence. The project team will identify gaps between current practices and best evidence, analyze barriers to implementing evidence-based guidelines, and develop strategies to facilitate their integration into clinical settings. The focus will also be on improving the knowledge and skills of pediatric nurses through targeted education and support. Ultimately, this initiative seeks to ensure the safety and effectiveness of gastric tube placement in the pediatric population, leading to better patient outcomes and higher standards of care.

DETAILED DESCRIPTION:
Enteral nutrition is the preferred method of nutritional support for children with gastrointestinal function, encompassing both oral and tube feeding approaches. Tube feeding involves delivering liquid food, water, and medications directly into the gastrointestinal tract through a feeding tube, making it a primary method of enteral nutrition. Compared to parenteral nutrition, enteral nutrition is more aligned with the body's physiological needs, helping to maintain the intestinal mucosal barrier, protect organ function, and regulate immune responses while being easier to initiate, cost-effective, and associated with a lower risk of infection.

In 2009, the American Society for Parenteral and Enteral Nutrition (ASPEN) published guidelines for enteral nutrition practices, which were updated in 2017. ASPEN also launched the Verification of Enteral Tube Location Project (NOVEL) in 2019, providing clear protocols for the placement of nasogastric tubes in children. Additionally, the European Society for Pediatric Gastroenterology, Hepatology, and Nutrition issued a position statement on nasoenteric feeding for children in 2019.

In China, pediatric clinical nutrition has developed more slowly, but pediatric tube feeding has received growing attention in recent years. The Chinese Society of Parenteral and Enteral Nutrition published clinical application guidelines for pediatric enteral and parenteral nutrition support in 2010, followed by neonatal nutrition support guidelines in 2013. However, there have been no recent updates or standardized procedures for pediatric tube feeding.

This study aims to synthesize the latest evidence on pediatric gastric tube placement and update healthcare professionals' knowledge in pediatric medical institutions, which also seeks to standardize tube placement techniques and apply best practices in clinical settings to enhance the safety and quality of care for children.

ELIGIBILITY:
Nurse Inclusion and Exclusion Criteria:

Inclusion:

* Nurses who hold a valid and legal nursing license.
* Nurses who have at least 1 year of clinical nursing experience in pediatric care.

Exclusion:

* Nurses who are on leave or not on duty.
* Nurses working in departments such as the operating room or intravenous compounding center, where nasogastric tube placement is not routinely performed.
* Nurses who are in training or on internships.

Pediatric Patient Inclusion and Exclusion Criteria:

Inclusion:

* Hospitalized children Aged 0-18 years.
* Scheduled for nasogastric tube placement.
* Parents or legal guardians have signed the informed consent form, agreeing to the child's participation in the study.

Exclusion:

* Presence of severe complications or unstable medical conditions.
* Nasogastric tube is intended for gastrointestinal decompression, drainage, or venting.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2750 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Compliance rate of gastric tube placement protocols among pediatric nursing staff | From baseline to the end of the 3 months implementation
  The total number of gastric tube placement procedures performed by nursing staff during the study period will be the denominator, while the number of procedures that comply with best evidence practice will be the numerator.

SECONDARY OUTCOMES:
Effects of evidence-based best practice interventions | From baseline to the end of the 3 months implementation
  First-attempt Success Rate of placement: The number of successful placements of the gastric tube at the correct position on the first attempt as the numerator, and the total number of placement attempts as the denominator.
  Adverse Event Rate: The number of adverse events occurring during placement as the numerator, and the total number of placement attempts as the denominator.
Pediatric nursing staff's personal knowledge level of gastric tube placement | From baseline to the end of the 3 months implementation
  "Nurses' knowledge of gastric tube placement questionnaire", a self-designed questionnaire was used to compare the correct rate before and after the intervention to test the intervention effect.

CONTACTS AND LOCATIONS:
Locations (22):
- China (22):
  - Children's Hospital of Fudan University, Shanghai, Minhang
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - Capital Center for Children's Health,Capital Medical University, Beijing
  - Peking University First Hospital, Beijing
  - Children's Hospital of Chongqing Medical University, Chongqing
  - Gansu Provincial Maternity and Child-care Hospital/Gansu Provincial Central Hospital, Gansu
  - Guangzhou Women and Children's Medical Center, Guangdong
  - Anhui Provincial Children's Hospital, Hefei
  - Henan Provincial People's Hospital, Henan
  - Hunan Children's Hospital, Hunan
  - The First Hospital of Jilin University, Jilin
  - Jinan Maternity and Child Health Care Hospital, Jinan
  - Kunming Children's Hospital, Kunming
  - Children's Hospital of Nanjing Medical University, Nanjing
  - Qingdao Women and Children's Hospital, Qingdao
  - Shengjing Hospital of China Medical University, Shenyang
  - Shenzhen Children's Hospital, Shenzhen
  - West China Second University Hospital, Sichuan University, Sichuan
  - Children's Hospital of Soochow University, Suzhou
  - The First People's Hospital of Urumqi （Urumqi Children's Hospital), Ürümqi
  - Tongji Hospital,Tongji Medical College of HUST, Wuhan
  - Children's hospital,Zhejiang University School of Medicine, Zhejiang

IPD SHARING:
Plan to Share IPD: No